CLINICAL TRIAL: NCT05711680
Title: INTERFACE: hIv patieNts TracER For clinicAl assistanCe and rEsearch During COVID 19 Epidemic: a Paradigm for Chronic Conditions
Brief Title: INTERFACE: hIv patieNts TracER For clinicAl assistanCe and rEsearch During COVID 19
Acronym: INTERFACE 3436
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3436
Record Dates: First submitted 2023-02-02; First posted 2023-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Device — To develop an e-health system to remotely monitor patients with chronic HIV infection and conduct early screening for COVID-19 through a telemonitoring, teleconsultation and periodic remote visit system.

SUMMARY:
The health emergency related to the SARS CoV2 pandemic has highlighted the problems of health management of patients at risk of COVID19 and with chronic diseases, suggesting the need for new methods of patient monitoring. Teleconsultation, and telemedicine in general, are applications that allow, at these times when access to hospitals is by definition limited, to monitor patients with chronic conditions who need regular and consistent care and monitoring. People living with HIV/AIDS (PLWHA) represent a paradigm of chronic patients on whom the development of e-health-based remote monitoring could have a significant impact in terms of maintaining an adequate standard of care. For these reasons, in a large teaching hospital we are planning the creation and use of an application to enable remote monitoring of PLWHA by combining the COVID19 prescreening system and chronicity monitoring.

ELIGIBILITY:
Inclusion criteria:

* Age of patients>18 years. Patients able to use apps and smart devices without caregivers or, if the patient is unable to use them, patients with caregivers able to use apps and smart devices.
* Able to provide informed consent

Exclusion criteria:

* Patients unable to use smart devices and apps without the presence of caregivers - Recent diagnosis of HIV infection (<3 months)
* Any unstable clinical condition requiring hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All PLWHA on antiretroviral therapy will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
A new model for patient follow-up | 1 year
  Develop an e-health system to remotely monitor patients with chronic HIV infection and conduct early screening for COVID-19 through a system of telemonitoring, teleconsultation and periodic remote visits.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST degli Ospedali Civili di Brescia, Brescia, BS
  - 3. Azienda Ospedaliera Universitaria Policlinico "San Martino" IRCCS di Genova, Genova, GE
  - Fondazione PoliclinicoAgostino Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No